CLINICAL TRIAL: NCT02549573
Title: Outpatient Physical Therapy Intervention in Subjects With Parkinson's DiseaseCurrently Using APOKYN®: A Phase IV Study of Outcome Assessments of Physical Therapy in Subjects in an "On" Versus "End-of-Dose-Off" Motor State
Brief Title: Outpatient Physical Therapy Intervention in Subjects With Parkinson's Disease Currently Using APOKYN®
Acronym: PERFORM
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Subject enrollment is unsatisfactory
Sponsor: MDD US Operations, LLC a subsidiary of Supernus Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Supernus Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: USWM-AP1-4002
Record Dates: First submitted 2015-09-09; First posted 2015-09-15 (Estimated); Results first posted 2018-01-12 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2017-12

CONDITIONS: Parkinson's Disease; Motor Symptoms
Keywords: Motor Symptoms; Parkinson's disease; Apokyn; Apomorphine; PD
MeSH Terms: conditions — Parkinson Disease | interventions — Apomorphine; Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Apokyn treatment before physical therapy (Active Comparator): APOKYN treatment before the PT Intervention Visit. Subjects in the "APO+" group will administer their usual dose of APOKYN at the PT clinic, as instructed by the Physical Therapist. These subjects will not take carbidopa/levodopa for at least 3 hours before or during the PT Intervention Visit.
  Interventions: Drug: APOKYN; Behavioral: Physical Therapy
- Apokyn treatment withheld before physical therapy (Other): APOKYN treatment withheld before the PT Intervention Visit. Subjects in the "APO-" group will not take carbidopa/levodopa and APOKYN for at least 3 hours before or during the PT Intervention Visit. No "rescue therapy" will be allowed during the PT. Intervention Visit. If the PT Intervention Visit needs to be stopped early, the Physical Therapist will record this along with a reason for the discontinuation.
  Interventions: Behavioral: Physical Therapy

INTERVENTIONS:
Drug: APOKYN — Subjects in the APOKYN+ group will administer his/her usual dose of APOKYN at the PT clinic, as instructed by the Physical Therapist. These subjects will not take carbidopa/levodopa for at least 3 hours before or during the PT Intervention Visit.
  Other Names: Apomorphine; APO
  Arms: Apokyn treatment before physical therapy
Behavioral: Physical Therapy — All subjects will participate in a standardized PT intervention
  Other Names: PT

SUMMARY:
To determine if PT intervention will be improved while in the "on" motor state vs. the "end-of-dose-off" motor state during the PT Intervention Visit in subjects with PD.

DETAILED DESCRIPTION:
Multicenter, outpatient trial to evaluate PT outcomes in subjects diagnosed with PD and currently using APOKYN. Those subjects who satisfy all eligibility criteria will be randomized to 2 treatment groups:

1. "APO+" (APOKYN treatment before the PT Intervention Visit) and;
2. "APO-" (APOKYN treatment withheld before the PT Intervention Visit).

The study will have:

* Baseline Assessment Visit(s) - 1 day at Investigator's clinic and PT clinic
* APOKYN Response Verification Visit - 1 day
* PT Intervention Visits - for 6 weeks
* End-of-study Assessment Visit(s) - 1 day at Investigator's clinic and PT clinic All subjects will participate in a standardized PT intervention. In both treatment groups, ALL subjects will arrive for the PT Intervention Visit in an "end-of-dose-off" motor state. The "end-of-dose-off" motor state will be achieved by the subject withholding his/her carbidopa/levodopa dose and APOKYN dose for at least 3 hours before the PT Intervention Visit. It is hypothesized that the outcome of PT will be improved when subjects are in the "on" motor state during PT Intervention visits compared with being in the "end-of-dose-off" motor state during PT Intervention visits.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and sign an Investigational Review Board (IRB)-approved written informed consent and privacy language (e.g., Health Insurance Portability and Accountability Act (HIPAA) authorization) as per national regulations before any study-related procedures are performed.
* Must have a diagnosis of idiopathic PD.
* Adult male or female 18 to 78 years of age, inclusive.
* Currently using APOKYN, per the Package Insert, for at least 4 weeks before Baseline Assessment Visit(s).
* Currently using carbidopa/levodopa therapy at a steady maintenance dose, representing a stable treatment regimen in the opinion of the Investigator, for at least 4 weeks before Baseline Assessment Visit(s).
* Able to walk 50 feet independently (cane permissible) at the Baseline Assessment Visit.
* Meet all of the following parameters to demonstrate an optimal response to APOKYN at the APOKYN Response Verification Visit: must be "on" in the opinion of the subject and investigator within 20 minutes after the APOKYN injection; and have a motor state improvement of >25% per the Movement Disorder Society (MDS)-UPDRS Motor Score (Part III), within 20 minutes after the APOKYN injection, as compared to pre-injection.
* Willing and able to comply with scheduled visits, treatment plan, other study-related procedures, and have available caregiver to provide transportation to clinic visits as needed.

Exclusion Criteria:

* Received PT targeting Parkinson's disease within 6 months before Baseline Assessment Visit(s).
* Received any investigational (i.e., unapproved) drug product within the last 30 days (or 5 half-lives, whichever is longer) before the Baseline Assessment Visit(s).
* Currently taking, or likely to need to take at any time during the course of the study, any 5HT3 antagonist (i.e., ondansetron, granisetron, dolasetron, palonosetron, alosetron).
* Currently on or likely to transition to the DUOPA (carbidopa and levodopa enteral suspension) during the course of the study.
* Has orthostatic hypotension (defined as >30 mmHg decrease in systolic blood pressure or >15 mmHg decrease in diastolic blood pressure within 2 minutes of standing from a supine position) at the Baseline Assessment Visit(s), or within 20 minutes following APOKYN injection at the APOKYN Verification Visit.
* Has a score of 24 or higher on the Modified Physical Performance Test (M-PPT).
* Has a score of 80% or higher on the Activities-specific Balance Confidence Scale (ABC).
* Has any significant current medical disorder, physical, or mental condition that would, in the Investigator's opinion, represent a hazard to the subject or prevent the subject from completing the study.
* Subjects with dementia, in the Investigator's opinion, or subjects with a Montreal Cognitive Assessment (MoCA) <18.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Pirner, MD, Study Director — US WorldMeds
Locations (12):
- United States (12):
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Loma Linda, California
  - Sunnyvale, California
  - Orlando, Florida
  - Foxborough, Massachusetts
  - Cleveland, Ohio
  - Tulsa, Oklahoma
  - Hershey, Pennsylvania
  - Austin, Texas
  - Kirkland, Washington
  - Tacoma, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Apokyn Treatment Before Physical Therapy | Apokyn Treatment Withheld Before Physical Therapy
Started | 6 | 7
Completed | 6 | 4
Not Completed | 0 | 3
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Apokyn Treatment Before Physical Therapy | Apokyn Treatment Withheld Before Physical Therapy | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 4 | 4 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 6 | 5 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 6 | 6 | 12
  Race: Hispanic | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Activities-specific Balance Confidence (ABC) Scale
Description: Scale from 0 to 100% where an increase in percent represents an improvement in balance confidence.
Time Frame: Baseline and after week 6
Population: The per protocol population included all subjects who completed at least 12 of the 18 physical therapy intervention visits within 6 weeks.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Apokyn Treatment Before Physical Therapy | Apokyn Treatment Withheld Before Physical Therapy
Number analyzed (Participants) | 6 | 4
percent change | 3.1 (8.70) | 15.2 (17.72)

2. Secondary Outcome: Change From Baseline in Movement Disorder Societies Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III (Motor Examination)
Description: MDS-UPDRS Part III is a sub-scale of MDS-UPDRS. Sub-scale scores range from 0 (best score possible) to 72 (worst score possible). A negative change from baseline represents an improvement in motor function.
Time Frame: Baseline and after week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apokyn Treatment Before Physical Therapy | Apokyn Treatment Withheld Before Physical Therapy
Number analyzed (Participants) | 6 | 4
units on a scale | -4.2 (10.01) | -0.8 (7.27)

3. Secondary Outcome: Change From Baseline in Modified Physical Performance Test (M-PPT)
Description: Investigator scale assessing 9 domains of physical functioning where total scores range from 0 to 28 with higher scores indicating better physical performance. A positive change from baseline represents an improvement in physical performance.
Time Frame: Baseline and after week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apokyn Treatment Before Physical Therapy | Apokyn Treatment Withheld Before Physical Therapy
Number analyzed (Participants) | 6 | 4
units on a scale | 3.8 (2.93) | 5.8 (4.11)

4. Secondary Outcome: Change From Baseline in Timed-Up-and-Go (TUG) Test
Description: Test captures the amount of time for a subject to get up from an arm chair, walk 3 meters, turn around, walk back to chair, and sit. A negative change from baseline represents an improvement of physical function.
Time Frame: Baseline and after week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Apokyn Treatment Before Physical Therapy | Apokyn Treatment Withheld Before Physical Therapy
Number analyzed (Participants) | 6 | 4
seconds | -4.0 (3.08) | 0.1 (2.13)

5. Secondary Outcome: Change From Baseline in 6-Minute Walk Test (6MWT)
Description: Objective performance based measure of functional exercise capacity that measures the distance a subject can cover on a 30 meter flat walking area over 6 minutes. A positive change from baseline represents an improvement in the distance walked (ft) in 6 minutes.
Time Frame: Baseline and after week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | Apokyn Treatment Before Physical Therapy | Apokyn Treatment Withheld Before Physical Therapy
Number analyzed (Participants) | 6 | 4
feet | 238.7 (191.88) | 315.3 (317.36)

6. Secondary Outcome: Change From Baseline in Montreal Cognitive Assessment (MoCA)
Description: The MoCA is a validated, 30-point test (sum of the 6 domains), with scores ranging from 0 (worst) to 30 (best). The test is designed to assess several cognitive domains, including visuospatial abilities (5 points), animal naming (3 points), attention (6 points), language (3 points), abstraction (2 points), delayed recall (5 points), and orientation to time and place (6 points). Total MoCA scores higher than 26 indicate normal cognitive function. A positive change from baseline represents an improvement in cognitive function.
Time Frame: Baseline and after week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apokyn Treatment Before Physical Therapy | Apokyn Treatment Withheld Before Physical Therapy
Number analyzed (Participants) | 6 | 4
units on a scale | 0.3 (1.21) | -0.3 (0.96)

7. Secondary Outcome: Change From Baseline in MDS-UPDRS Part I A
Description: MDS-UPDRS Part I A is a sub-scale of MDS-UPDRS. Sub-scale scores range from 0 (best score possible) to 24 (worst score possible). A negative change from baseline represents an improvement in non-motor experiences of daily living (investigator rated).
Time Frame: Baseline and after week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apokyn Treatment Before Physical Therapy | Apokyn Treatment Withheld Before Physical Therapy
Number analyzed (Participants) | 6 | 4
units on a scale | -0.3 (1.21) | -2.3 (2.50)

8. Secondary Outcome: Number of Participants in Each Category of Clinical Global Impression of Change (CGI-C)
Description: Investigator's impression of change in the subject's symptoms from baseline assessment visit to end of study assessment, on a 7-point scale ranging from very much improved to very much worse.
Time Frame: After week 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Apokyn Treatment Before Physical Therapy | Apokyn Treatment Withheld Before Physical Therapy
Number analyzed (Participants) | 6 | 4
Participants
  Minimally Improved | 2 | 2
  Much Improved | 3 | 2
  Very Much Improved | 1 | 0

9. Other Pre Specified Outcome: Change From Baseline in Parkinson's Disease Questionnaire (PDQ-39)
Description: PDQ-39 is a scale measuring subject reported aspects of functioning and well-being. Each of the 39 items is rated using a 5-points Likert scale, with 0 for never having difficulties/problems and 4 for all always having difficulties/problems. The total score is the sum of the 39 items, with a minimum score of 0 and a maximum score of 156. A negative change from baseline represents an improvement in functioning and well-being.
Time Frame: Baseline and after week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apokyn Treatment Before Physical Therapy | Apokyn Treatment Withheld Before Physical Therapy
Number analyzed (Participants) | 6 | 4
units on a scale | 4.8 (5.71) | -8.8 (8.88)

10. Other Pre Specified Outcome: Change From Baseline in Parkinson's Fatigue Scale (PFS-16)
Description: PFS-16 is a subject-reported scale evaluating the physical effects of fatigue and its impact on daily function, with a minimum score of 16 and a maximum score of 80. Ratings are based on feelings and experiences over the prior 2 weeks, with scoring ranging from 1 (strongly disagree) to 5 (strongly agree), where lower scores are associated with less fatigue and higher scores are associated with greater fatigue.
  A negative change from baseline represents an improvement in the physical effects of fatigue and the impact on daily function. .
Time Frame: Baseline and after week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apokyn Treatment Before Physical Therapy | Apokyn Treatment Withheld Before Physical Therapy
Number analyzed (Participants) | 6 | 4
units on a scale | -3.5 (10.27) | -8.3 (7.72)

11. Other Pre Specified Outcome: Hospital Anxiety and Depression Scale - Change From Baseline in Anxiety
Description: The Hospital Anxiety and Depression Scale is a 14-item Investigator-rated scale designed to determine levels of anxiety and depression in people with physical health problems. Seven items relate to anxiety and 7 items related to depression, where the scale ranges from 0 (best score possible) to 21 (worst score possible). A negative change from baseline represents a decrease in anxiety.
Time Frame: Baseline and after week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apokyn Treatment Before Physical Therapy | Apokyn Treatment Withheld Before Physical Therapy
Number analyzed (Participants) | 6 | 4
units on a scale | 0.3 (2.73) | 1.0 (2.83)

12. Other Pre Specified Outcome: Number of Participants in Each Category of Patient Global Impression of Change (PGI-C)
Description: Self reported (caregiver, if applicable) impression of change in the subject's symptoms from baseline assessment visit to end of study assessment, on a 7-point scale ranging from much improved to very much worse.
Time Frame: After week 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Apokyn Treatment Before Physical Therapy | Apokyn Treatment Withheld Before Physical Therapy
Number analyzed (Participants) | 6 | 4
Participants
  No Change | 1 | 0
  Minimally Improved | 1 | 3
  Much Improved | 2 | 1
  Very Much Improved | 1 | 0
  Data Not Collected | 1 | 0

13. Other Pre Specified Outcome: Change From Baseline in Number of Falls as Reported by the Subject in the Past 1 Week
Description: Subject reported number of falls. A negative change from baseline represents a decrease in the frequency of falls.
Time Frame: Baseline and after week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of falls reported
Arm/Group | Apokyn Treatment Before Physical Therapy | Apokyn Treatment Withheld Before Physical Therapy
Number analyzed (Participants) | 6 | 4
number of falls reported | 0 (0) | -1.0 (0.82)

14. Secondary Outcome: Change From Baseline in MDS-UPDRS Part II
Description: MDS-UPDRS Part II is a sub-scale of MDS-UPDRS. Sub-scale scores range from 0 (best score possible) to 52 (worst score possible). A negative change from baseline represents an improvement in motor experience of daily living.
Time Frame: Baseline and after week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apokyn Treatment Before Physical Therapy | Apokyn Treatment Withheld Before Physical Therapy
Number analyzed (Participants) | 6 | 4
units on a scale | -0.7 (3.01) | -1.3 (2.87)

15. Secondary Outcome: Change From Baseline in MDS-UPDRS Part IV
Description: MDS-UPDRS Part IV is a sub-scale of MDS-UPDRS. Sub-scale scores range from 0 (best score possible) to 24 (worst score possible). A negative change from baseline represents fewer motor complications.
Time Frame: Baseline and after week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apokyn Treatment Before Physical Therapy | Apokyn Treatment Withheld Before Physical Therapy
Number analyzed (Participants) | 6 | 4
units on a scale | 1.2 (1.47) | 0 (1.63)

16. Secondary Outcome: Change From Baseline in MDS-UPDRS Part I B
Description: MDS-UPDRS Part I B is a sub-scale of MDS-UPDRS. Sub-scale scores range from 0 (best score possible) to 28 (worst score possible). A negative change from baseline represents an improvement in non-motor experiences of daily living (subject rated).
Time Frame: Baseline and after week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apokyn Treatment Before Physical Therapy | Apokyn Treatment Withheld Before Physical Therapy
Number analyzed (Participants) | 6 | 4
units on a scale | 1.0 (4.43) | -0.8 (3.50)

17. Secondary Outcome: Change From Baseline in Clinical Global Impression of Severity (CGI-S)
Description: Investigator's impression of the severity of the subject's illness on a 7-point scale ranging from normal (1) to among the most extremely ill subjects (7). A negative change from baseline represents a decrease in the severity of the subject's illness.
Time Frame: Baseline and after week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apokyn Treatment Before Physical Therapy | Apokyn Treatment Withheld Before Physical Therapy
Number analyzed (Participants) | 6 | 4
units on a scale | -0.7 (0.82) | 0 (0.82)

18. Other Pre Specified Outcome: Change From Baseline in Patient Global Impression of Severity (PGI-S)
Description: Self reported (caregiver, if applicable) impression of the severity of the subject's illness on a 7-point scale ranging from normal (1) to among the most extremely ill subjects (7). A negative change from baseline represents a decrease in the severity of the subject's illness.
Time Frame: Baseline and after week 6
Population: The per protocol population included all subjects who completed at least 12 of the 18 physical therapy intervention visits within 6 weeks. One subject in APO+ group did not have an end of study assessment for PGI-S.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apokyn Treatment Before Physical Therapy | Apokyn Treatment Withheld Before Physical Therapy
Number analyzed (Participants) | 5 | 4
units on a scale | 0.4 (1.14) | 0 (0.82)

19. Other Pre Specified Outcome: Hospital Anxiety and Depression Scale - Change From Baseline in Depression
Description: The Hospital Anxiety and Depression Scale is a 14-item Investigator-rated scale designed to determine levels of anxiety and depression in people with physical health problems. Seven items relate to anxiety and 7 items related to depression, where the scale ranges from 0 (best score possible) to 21 (worst score possible). A negative change from baseline represents a decrease in depression.
Time Frame: Baseline and after week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apokyn Treatment Before Physical Therapy | Apokyn Treatment Withheld Before Physical Therapy
Number analyzed (Participants) | 6 | 4
units on a scale | -0.5 (2.88) | -1.0 (2.94)

ADVERSE EVENTS:
Groups:
- Apokyn Treatment Withheld Before Physical Therapy: APOKYN treatment withheld before the PT Intervention Visit. Subjects in the "APO-" group will not take carbidopa/levodopa and APOKYN for at least 3 hours before or during the PT Intervention Visit. No "rescue therapy" will be allowed during the PT Intervention Visit. If the PT Intervention Visit needs to be stopped early, the Physical Therapist will record this along with a reason for the discontinuation.
  Physical Therapy: All subjects will participate in a standardized PT intervention
Arm/Group | Apokyn Treatment Before Physical Therapy | Apokyn Treatment Withheld Before Physical Therapy
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/7
Other Adverse Events (participants affected / at risk) | 0/6 | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apokyn Treatment Before Physical Therapy (N=6) | Apokyn Treatment Withheld Before Physical Therapy (N=7)
Accelerated Hypertension (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Recruitment challenges (primarily due to standardized physical therapy requirements within sites) led to trial termination. The small number of subjects resulted in statistically unreliable results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the first right, within 9 months following the later to occur 1) close out meeting or 2) Sponsor possessing all data, to publish the lead paper. Following the foregoing, Institution has the right to publish the results provided the Institution provides a Publications Committee, which includes the Sponsor, with a draft at least 30 days before submission. At Sponsor's request, Institution shall withhold publication for 45 days to allow filing of a patent application.